CLINICAL TRIAL: NCT00390715
Title: Prospective Study of the Value of the Cytogenetic and of the Monitoring of the Minimal Residual Disease
Brief Title: Treatment of Acute Myeloblastic Leukemia in Younger Patients
Status: Completed | Type: Observational
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Pethema, pethema
Other Study IDs: AML99<=65 años
Record Dates: First submitted 2006-10-18; First posted 2006-10-20 (Estimated); Last update posted 2010-03-15 (Estimated); Status verified 2010-03

CONDITIONS: Acute Myeloblastic Leukemia
Keywords: Acute Myeloblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: chemotherapy

SUMMARY:
study of the value of the cytogenetics and the monitoring of the residual minimum disease in the standard treatment of acute myeloblastic leukemia.

DETAILED DESCRIPTION:
The treatment scheme is purely welfare and therefore it does not require any approval of ethical committees for his application. It gathers the basic ideas of the present treatment of the AML, with optional induction according to preference of each center with daunorubicin or Idarubicin (x3) associated to AraC (x7). The patients who reach CR consolidate with an identical cycle to the used one in the induction. Later (if pte has identical donor HLA, and as much it as their doctors has preference by this option) receive allogenic transplant. The other patients who reach CR receive two intensifications, one that AraC to intermediate dose contains and another one with autologous transplant, previous preparation with Busulfán, Etoposide and AraC. Later all antileucemic treatment is suspended until possible relapse. This scheme of treatment is accompanied by a valuation of the quality of the CR with traditional morphology, Immunocytometry and molecular genetic study and of a pursuit of residual minimum disease (EMR) using the same techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age< or =65 years.
* ECOG<=3.
* AML of new diagnose.
* Consent for chemotherapy.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AML of new diagnose, no treated previously
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 1999-01; Primary Completion 2007-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diaz Mediavilla Joaquin, Dr, Study Chair — Hospital Clínico Universitario San Carlos
Locations (42):
- Spain (42):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital Clínic, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona, Barcelona
  - Hospital vall d'Hebrón, Barcelona, Barcelona
  - Hospital Valle Hebrón-Materno Infantil, Barcelona, Barcelona
  - Xarxa assistencial de Manresa, Manresa, Barcelona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital general de Castellón, Castelló, Castellón
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Complejo Hospitalario Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hospital Juan Canalejo, A Coruña, La Coruña
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - Hospital Doce de Octubre, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid, Madrid
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Hospital General Universitario Morales Meseguer., Murcia, Murcia
  - . Hospital Clínico Universitario Virgen de la Victoria, Málaga, Málaga
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Oviedo
  - Hospital Son Dureta, Palma de Mallorca, Palma de Mallorca
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona, Tarragona
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Hospital Clínic, Valencia, Valencia
  - Hospital La Fe, Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia, Valencia
  - Complejo Hospitalario Xeral-Cies, Vigo, Vigo
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza
  - Complejo Hospitalario de Cáceres, Cáceres
  - Area Hospitalaria Juan Ramón Jimenez, Huelva
  - Hospital general de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Virgen Blanca de León, León
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital General de Segovia, Segovia
  - Hospital Txagorritxu, Vitoria-Gasteiz

REFERENCES:
- See also: Spanish association of Haematology — http://www.aehh.org